CLINICAL TRIAL: NCT00572026
Title: Enhancing ADHD Driving Performance With Stimulant Medication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Daniel J. Cox, PhD, University of virginia
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 12189
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention deficit; Hyperactivity; Attention deficit hyperactivity disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Daytrana
  Interventions: Drug: Methylphenidate Transdermal System
- 2 (No Intervention): No treatment for ADHD

INTERVENTIONS:
Drug: Methylphenidate Transdermal System — Daytrana wear time up to 15 hours
  Other Names: Brand name = Daytrana
  Arms: 1

SUMMARY:
Among children, attention-deficit/hyperactivity disorder (ADHD) is associated with an increased risk for accidents, especially bicycle and pedestrian (Leibson 2001; Jensen 1988; DiScala 1998). Anywhere from 40% to 80% of children diagnosed with ADHD continue to display symptoms of the disorder into adolescence(Barkley 1990; Gittelman 1985). Adolescents with ADHD are also at an increased risk for driving-related accidents, being 2 to 4 times more likely to experience a motor vehicle accident (Barkley 1993; Barkley 1996; Cox 2000), 4 times as likely to be at fault in the accident (Barkley 1993), and over 3 times more likely to incur associated injuries as a result of the accident(Murphy 1996).

Stimulant treatment with immediate-release methylphenidate (IR MPH) has been demonstrated to improve driving performance in adolescents with ADHD.

Hypothesis to be Tested:

* Main study: Just as stimulant medication improves simulation and on-road driving performance of ADHD teenagers, it is hypothesized that stimulant medication will improve routine driving performance.
* Substudy - Extended wear (15 hours) of Daytrana will lead to safer driving late in the evening (22:00 and 01:00), when the most dangerous driving mishaps are most likely to occur, and the next morning at 09:00.

DETAILED DESCRIPTION:
Driving collisions are the leading cause of death among adolescents, accounting for 15 teenage deaths per day in the United States. (National Highway Traffic Safety Administration 2003). Driving fatalities are significantly more likely to occur when distracting teenage passengers are in the automobile(Insurance Institute for Highway Safety 2000). Fatalities are also more likely to occur in the evenings, on the weekends, and during the summer months (National Center for Statistics and Analysis 2005).

Among children, attention-deficit/hyperactivity disorder (ADHD) is associated with an increased risk for accidents, especially bicycle and pedestrian (Leibson 2001; Jensen 1988; DiScala 1998). Anywhere from 40% to 80% of children diagnosed with ADHD continue to display symptoms of the disorder into adolescence(Barkley 1990; Gittelman 1985). Adolescents with ADHD are also at an increased risk for driving-related accidents, being 2 to 4 times more likely to experience a motor vehicle accident (Barkley 1993; Barkley 1996; Cox 2000), 4 times as likely to be at fault in the accident (Barkley 1993), and over 3 times more likely to incur associated injuries as a result of the accident(Murphy 1996).

Stimulant treatment with immediate-release methylphenidate (IR MPH) has been demonstrated to improve driving performance in adolescents with ADHD. Simulated driving performance was assessed 1.5 to 2 hours post-dose in a double-blind, crossover study comparing the effects of one 10-mg dose of immediate-release methylphenidate (IR MPH) with placebo in male subjects with ADHD (aged 19-25 years) to that of matched controls without ADHD(Cox 2000). When placebo was administered to both groups, ADHD-diagnosed participants demonstrated significantly poorer driving scores than did controls (P<0.05); however, 1.5 hours after the administration of IR MPH, the driving performance of the ADHD-diagnosed group significantly improved (P<0.05) and was equivalent to that of the control group.

To determine whether the difference in the pharmacokinetic profiles of IR and extended-release MPH formulations influenced driving performance throughout the day, a study was conducted to compare IR MPH dosed 3 times daily (tid) with once-daily, OROS® MPH (CONCERTA®) (Cox 2004a). OROS MPH delivers MPH via an osmotic pump to produce an ascending profile with duration of treatment effect through 12 hours(Swanson 2003). Once-daily dosing of OROS MPH is similar to IR MPH dosed tid and minimizes the fluctuations in peak and trough plasma concentrations associated with MPH dosed tid(Swanson 2003). Therefore, in this crossover study design, OROS MPH was administered at 8:00 AM, and IR MPH was administered tid at 8:00 AM, 12:00 PM, and 4:00 PM. The driving performance of adolescents with ADHD aged 16 to 19 years was assessed using a driving simulator at 2:00, 5:00, 8:00 and 11:00 PM. When subjects were administered IR MPH, simulated driving performance worsened by a factor of 5 at 8:00 PM and 11:00 PM, but driving performance in subjects receiving OROS MPH remained stable from 2:00 PM to 11:00 PM. Not only was driving performance significantly better in subjects receiving OROS MPH (P<0.001), but subjects treated with OROS MPH demonstrated significantly less variability in driving performance (P<0.001).

In a subsequent study to compare driving skills in subjects receiving and not receiving medication, adolescents with ADHD drove their own car on a standard road course after either taking OROS MPH at 8:00 AM or receiving no medication. (Cox 2004b) Raters, who were blinded to the medication condition, observed significantly fewer inattentive driving errors in adolescents taking OROS MPH (P<0.01). The study demonstrated that reduction in inattentive errors was positively correlated (r=0.60, P<0.01) with mg/kg dosing of OROS MPH.

Given the evidence that stimulant therapy with MPH improves driving performance and that once-daily OROS MPH improves driving performance and is more effective in the evenings compared with the IR formulation, we recently studied the effects of 2 long-acting stimulant formulations-once-daily OROS MPH and mixed amphetamine salts extended release (se AMPH ER, ADDERALL® XR)-on simulated driving performance in adolescents with ADHD to compare how each affected adolescent driving performance. This study indicated that medication improved driving performance and neuropsychological functioning relative to placebo, and that generally OROS MPH (Concerta) led to greater improvement. However, individual differences were such that a minority of subjects performed better when taking se AMPH ER (Adderall XR).

ELIGIBILITY:
Inclusion Criteria:

* ADHD diagnosis
* Valid driver's license
* Not taking any medication for their ADHD
* Have access to a car of which they are the primary driver
* Have a history of approximately two driving collisions or citations
* Have a history of responsiveness to methylphenidate

Exclusion Criteria:

* Older than 25 years of age
* Bi-polar disease
* Psychosis
* Satisfy the DSM IV criteria of active depressive or anxiety disorders
* Have any medical condition that might impair driving or be contra-indicated for the use of methylphenidate
* Pregnant or intending to get pregnant for the duration of the study,breastfeeding or intending to breastfeed for the duration of the study
* Have skin allergies or skin condition that could be exacerbated by wearing the medication patch
* Have documented allergy, hypersensitivity, or intolerance to methylphenidate
* Have documented hypersensitivity to the Daytrana® adhesive backing
* Have (history of):

  * seizures (except febrile seizure in infancy)
  * liver or renal disease
  * glaucoma
  * chronic skin conditions or contact sensitivities
  * current symptoms suggestive of cardiac disease
  * cardiovascular disease, e.g.
  * structural cardiac abnormalities
  * cardiac Arrythmias
  * cardiomyopathy
  * hypertension
  * reported ECG abnormality
  * vocal tics, motor tics, Tourettes Disorder or family history of Tourettes
* Have a current diagnosis of

  * Psychosis
  * Bi-polar disease
  * Anxiety disorder
  * Substance Use Disorder/Substance Abuse Disorder

Substudy: In addition to the above requirements, in order to participate in the substudy, participants must be capable of driving the simulator without experiencing simulation sickness

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Video recording of driving mishaps | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Cox, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States